CLINICAL TRIAL: NCT06995937
Title: An Open Road Driving Performance Task to Examine Long-term Medical Marijuana Use and Prescription Opioid Positivity in Adults 50 and Older
Brief Title: Medical Marijuana and Open Road Driving Task
Acronym: ROADACE
Status: Recruiting | Type: Observational
Sponsor: Florida State University (Other)
Collaborators: University of Florida (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Nicole Ennis, Principal Investigator, Florida State University
Other Study IDs: STUDY00005560; 1R01DA057965 (NIH)
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Medical Cannabis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical Marijuana Use (MMG): Individuals aged 50 and older who report medical marijuana use >12 months daily or most days of the week
- No Marijuana Exposure (NMG): Individuals aged 50 and older who report no marijuana exposure past 10 years (race-sex matched to MMG group).

SUMMARY:
Medical marijuana use among adults 50 and older has more than doubled in the past decade with exponential increases projected in this demographic by 2050, and prescription opioids are one of the most common treatments for pain management in this population. To date, no studies systematically assess driving performance in a rigorous and ecologically valid manner accounting for long-term medical marijuana use and/or the combined effect of prescription opioid use in adults 50 and older who endorse chronic or severe non-malignant pain. Further, studies examining how older adults self-regulate prescription medication use and driving behavior is limited, with none rigorously examining medical marijuana.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 and older who endorse chronic or severe non-malignant pain
* Resident of Florida with an active and valid Florida Drivers License
* Can communicate in English
* Willing and able to complete study procedures
* Have active medical marijuana card for >12 months issued by the state of Florida (MMG group) OR are race-sex match who has not used marijuana in the past 10 years with no history of daily use (NMG group)

Exclusion Criteria:

* Have active psychosis
* Have lost or revoked driving privileges
* Score of below the cut 24 (out of 30) on the Montreal Cognitive Assessment (MoCA)
* Are a control participant who urine test positive for marijuana use and/or reports any marijuana use in past 10 years

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Biological men and women in the state of Florida aged 50 and older
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2029-01-30 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Sum of Maneuvers Score (SMS) | One Day
  A standardized score sheet with a total of 49 driving maneuvers and eight types of possible driving errors is used by the Certified Driver Rehabilitation Specialist while the participant is driving. The driving errors are lane maintenance errors, speed regulation errors, adjustment-to-stimuli errors, yielding errors, signaling errors, vehicle positioning errors, visual scanning, and gap acceptance errors. For each maneuver, a maximum score of 3 is given if no errors are committed. At the end of the driving course, the sum of the points attained is computed as the sum of maneuvers score (SMS) ranging from 0 to 147, with 147 indicating a perfect driving score (zero errors).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Florida State University, Center for Translational Behavioral Science, Tallahassee, Florida

REFERENCES:
- [Derived] Ennis N, Classen S. An Open-Road Driving Performance Task to Examine Long-Term Medical Marijuana Use and Prescription Opioid Positivity Among Adults Aged 50 Years and Older: Protocol for an Observational Trial. JMIR Res Protoc. 2025 Nov 28;14:e77944. doi: 10.2196/77944. PMID 41313623